CLINICAL TRIAL: NCT04270448
Title: Effects of Feedback on Learning of a Motor Sequence Task
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Jill Stewart, PT, PhD, Associate Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00095119
Record Dates: First submitted 2020-02-04; First posted 2020-02-17 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Adult
Keywords: Motor learning; Feedback

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Practice of a joystick based motor sequence task. Participants receive feedback that they have completed the practice trials in that block of practice.
  Interventions: Behavioral: Motor Sequence Task
- Performance Feedback (Experimental): Practice of a joystick based motor sequence task. Participants receive feedback on their response time to complete the trials in the practice block.
  Interventions: Behavioral: Motor Sequence Task
- Performance plus Positive Feedback (Experimental): Practice of a joystick based motor sequence task. Participants receive feedback on their response time to complete the trials in the practice block plus positive social comparative feedback.
  Interventions: Behavioral: Motor Sequence Task

INTERVENTIONS:
Behavioral: Motor Sequence Task — Participants will be seated at a laptop with the right hand on a standard joystick. The movement of the joystick will move a cursor on the computer screen. Targets will appear on the laptop screen as a circle in one of twelve spatially distinct locations. The learner must move the joystick "cursor" to inside the target before the next target will appear.

SUMMARY:
Feedback delivered during motor practice can help promote motor skill learning and promote confidence. However, the optimal way to provide feedback to promote learning and confidence is unknown. This project will study how the feedback that is provided during practice of a movement skill can help people learn and build confidence. The investigators will measure motor skill performance and confidence before and after a session of motor practice.

DETAILED DESCRIPTION:
Feedback may be a useful tool to optimize motor learning during practice. For example, feedback during practice that indicates the learner is performing above average (i.e. positive social comparative feedback) enhances motor skill learning and self-efficacy in healthy adults. While this type of feedback is hypothesized to promote learning in some tasks, no studies have examined whether positive social comparative feedback during practice promotes motor learning in a traditional motor sequence task. Therefore, the aim of the proposed project is to investigate the effect of positive social comparative feedback on the learning of a joystick-based motor sequence task in healthy adults. The study aims to recruit 60 participants who will be randomized into 1 of 3 feedback groups (control group, performance feedback, and performance plus positive feedback). Participants will practice a motor sequence task on a single day and then return for retention performance testing about 24 hours later. Changes in performance (response time to complete a sequence) and self-efficacy will be measured from baseline to 24 hours later at retention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 40 years
* Right-hand dominant

Exclusion Criteria:

* Medical diagnosis or medication that affects dopamine (e.g. dopamine reuptake inhibitors)
* musculoskeletal issues that limit upper extremity movement

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Response Time | Change from baseline to retention at 24 hours
  Time to complete one sequence
Task Confidence | Change from baseline to retention at 24 hours
  Self-reported confidence in ability to complete a sequence in a given time on a scale of 0 to 10 with a 10 equating to higher confidence

SECONDARY OUTCOMES:
Peak Velocity | Change from baseline to retention at 24 hours
  Average speed to capture a target within a sequence
Peak Velocity | Change from baseline to immediately after practice
  Average speed to capture a target within a sequence
Total Path Distance | Change from baseline to retention at 24 hours
  Total distance traveled to complete one sequence
Total Path Distance | Change from baseline to immediately after practice
  Total distance traveled to complete one sequence
Time to Peak Velocity | Change from baseline to retention at 24 hours
  Mean time to peak velocity for movement to a target within a sequence
Time to Peak Velocity | Change from baseline to immediately after practice
  Mean time to peak velocity for movement to a target within a sequence
Perceived Competence | Change from baseline to retention at 24 hours
  Mean score on the Perceived Competence subscale of the Intrinsic Motivation Inventory where each item ranges from 0 to 7 with a higher value equating to higher competence
Perceived Competence | Change from baseline to immediately after practice
  Mean score on the Perceived Competence subscale of the Intrinsic Motivation Inventory where each item ranges from 0 to 7 with a higher value equating to higher competence
Perceived Interest/Enjoyment | Change from baseline to retention at 24 hours
  Mean score on the Interest/Enjoyment subscale of the Intrinsic Motivation Inventory where each item ranges from 0 to 7 with a higher value equating to higher enjoyment
Perceived Interest/Enjoyment | Change from baseline to immediately after practice
  Mean score on the Interest/Enjoyment subscale of the Intrinsic Motivation Inventory where each item ranges from 0 to 7 with a higher value equating to higher enjoyment
Positive Affect | Change from baseline to retention at 24 hours
  Total score for general positive affect on the Positive and Negative Affect Scale with a range from 10 to 50 with higher scores equating to higher positive affect
Positive Affect | Change from baseline to immediately after practice
  Total score for general positive affect on the Positive and Negative Affect Scale with a range from 10 to 50 with higher scores equating to higher positive affect
Response Time | Change from baseline to immediately after practice
  Time to complete one sequence
Task Confidence | Change from baseline to immediately after practice
  Self-reported confidence in ability to complete a sequence in a given time on a scale of 0 to 10 with a 10 equating to higher confidence

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available per reasonable request to the principal investigator 1 year after study completion.
Supporting Information: Study Protocol
Time Frame: 1 year after study completion